CLINICAL TRIAL: NCT06243588
Title: Identification of Prognostic Factors and Role of Radiotherapy in Patients With Ewing Sarcoma
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: ProEwing
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: patients treated at Rizzoli Institute from 1991 to 2021.
  Interventions: Other: clinical records review

INTERVENTIONS:
Other: clinical records review — review the medical records, radiological imaging, and histological data of these patients

SUMMARY:
assess whether there is a correlation between some factors (age, sex, tumor volume, tumor site, chemotherapy-induced necrosis, radiation and biomarkers) and overall survival (OS) and relapse-free survival (RFS) in patients with Ewing sarcoma.

Identification of reliable prognostic factors could help to identify high-risk patients, which may require a different treatment and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients treated at Rizzoli Orthopaedic Institute between 01/01/1991 and 31/12/2021
* Age ≥ 2 years
* Diagnosis of Ewing Sarcoma
* Patients with available clinical and imaging data

Exclusion Criteria:

* At least one inclusion criterion not met

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients treated at Rizzoli Orthopaedic Institute between 01/01/1991 and 31/12/2021
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation | At baseline (Day 0)
  Correlation between some factors (age, sex, tumor volume, tumor site, chemotherapy-induced necrosis, radiation and biomarkers) and overall survival (OS) and relapse-free survival (RFS) in patients with Ewing sarcoma.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Itituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grunewald TGP, Cidre-Aranaz F, Surdez D, Tomazou EM, de Alava E, Kovar H, Sorensen PH, Delattre O, Dirksen U. Ewing sarcoma. Nat Rev Dis Primers. 2018 Jul 5;4(1):5. doi: 10.1038/s41572-018-0003-x. PMID 29977059
- [Result] Pressman BD, Tourje EJ, Thompson JR. An early CT sign of ischemic infarction: increased density in a cerebral artery. AJR Am J Roentgenol. 1987 Sep;149(3):583-6. doi: 10.2214/ajr.149.3.583. PMID 3497548